CLINICAL TRIAL: NCT03203460
Title: A Phase II Randomized Controlled Trial of Exercise in Prostate Cancer Patients Undergoing Active Surveillance
Brief Title: Exercise During Active Surveillance for Prostate Cancer
Acronym: ERASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-17-0248
Record Dates: First submitted 2017-06-20; First posted 2017-06-29 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Exercise; High-Intensity Interval Training; Randomized Controlled Trial
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group assignment for the primary outcome of natural killer cell cytotoxic activity and the secondary outcomes of other circulating biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Supervised high-intensity aerobic interval training (HIIT) during active surveillance
  Interventions: Behavioral: High-intensity aerobic interval training (HIIT)
- Usual Care Group (No Intervention): The usual care group will be provided with standard active surveillance medical care.

INTERVENTIONS:
Behavioral: High-intensity aerobic interval training (HIIT) — A 12-week, supervised, HIIT aerobic exercise program consisting of alternating vigorous- and low-intensity intervals
  Arms: Exercise Group

SUMMARY:
The broad goal of the Exercise During Active Surveillance for Prostate Cancer (ERASE) trial is to examine the effects of exercise in prostate cancer patients undergoing active surveillance.

DETAILED DESCRIPTION:
The ERASE Trial will be a phase II randomized controlled trial. A total of 66 men with low- or intermediate-grade clinically localized prostate cancer undergoing active surveillance will be randomized to either a 12-week of supervised high-intensity aerobic interval training or usual care. The primary outcome will be peak oxygen consumption (VO2peak) as a measure of physical fitness. The secondary outcomes include tumour-related biomarkers, fear of cancer progression, quality of life, and psychological distress. Exploratory outcomes will include indicators of cancer progression including prostate-specific antigen. Based on this sample size, our study has 80% power with a two-tailed alpha <0.05 to detect a clinically meaningful effect of 3.5 ml/kg/min on our primary outcome of VO2max. This power will also be sufficient for detecting differences in our secondary biomarkers and patient-reported outcomes if the effects are at least moderate (i.e., a standardized effect size of d=0.60).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* diagnosed with low or favorable intermediate grade localized PCa defined as PSA less than 10, Gleason Score 3+3 or 3+4 with low volume, and digital rectal examination (DRE) of T1C or T2A
* initiating or continuing active surveillance with no plans for treatment for prostate cancer in the next 6 months (e.g., radical prostatectomy, radiotherapy, or androgen deprivation therapy)
* screened for medical clearance for exercise testing and participation in vigorous aerobic exercise
* residing in a commutable area near Edmonton, Alberta
* willing to commute to the Behavioural Medicine Fitness Centre three times per week to attend a 12-week supervised high-intensity aerobic interval exercise program

Exclusion Criteria:

* having comorbidities or uncontrolled medical conditions that their referred clinicians indicate as inappropriate to participate in exercise (e.g., known cardiac disease or uncontrolled hypertension)
* having contraindications for cardiopulmonary stress and/or physical fitness tests
* currently participating in a structured, vigorous exercise program.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Changes of Peak Oxygen Consumption (VO2peak) | At baseline and 12-week (postintervention)
  VO2peak is a measure of cardiopulmonary fitness and a powerful surrogate outcome for cancer-specific and overall survival. VO2peak will be defined as the highest oxygen-uptake value recorded during the test and quantified where participants reach a plateau in oxygen consumption, which will be expressed as relative to body mass (i.e., ml O2·kg-1·min-1).

SECONDARY OUTCOMES:
Changes of Natural Killer Cell Cytotoxic Activity (NKCA) and Counts | At baseline and 12-week (postintervention)
  NKCA significantly contributes to the regulation of tumour suppression in response to exercise and it has been demonstrated to have a diagnostic value in patients with cancer. NK cell activities are assessed using blood analysis as the total number of circulating NK cells and their cytotoxic activity. NK cell counts and NKCA will be measured using the phenotypic markers of NK cells (CD3-CD16+CD56+). NKCA will be expressed as the percentage of target cells killed by a sample of 100,000 peripheral blood mononuclear cells at the effector-to-target ratios of 5:1, 20:1, 40:1, and 100:1.
Changes of Immune-Related Phenotype | At baseline and 12-week (postintervention)
  Immune-related phenotypic markers, including CD3, CD16, CD56, and CD107 (on the frozen) and CD4, CD8, CD20, CD25, CD11, CD45RA, CD45RO, CD16, CD56, CD107 activation (fresh on whole blood), will be assessed using blood samples.
Changes of Prostate-Specific Antigen (PSA) | At baseline, 12-week (postintervention)
  PSA will be assessed using blood samples.
Changes of Complete Blood Count with Differential (CBCD) | At baseline and 12-week (postintervention)
  CBCD, including RBC, WBC, HGB, HCT, PLT, LYMPH, BASO, EOS, MONO, NEUT, will be assessed using blood samples.
Changes of Insulin | At baseline and 12-week (postintervention)
  Fasting insulin levels will be assessed using blood samples.
Changes of Fasting Glucose | At Baseline and 12-week postintervention
  Fasting glucose levels will be assessed using blood samples.
Changes of HbA1c | At Baseline and 12-week postintervention
  HbA1c will be assessed using using blood samples.
Changes of Insulin-like Growth Factor (IGF)-axis | At baseline and 12-week (postintervention)
  IGF-axis, including circulating IGF-1 and IGF binding protein(IGFBP)-3, will be assessed using blood samples.
Changes of Pro-Inflammatory Cytokines | At baseline and 12-week (postintervention)
  Pro-inflammatory cytokines, including IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, and TNF-α, will be assessed.
Changes of High-Sensitivity C-Reactive Protein (hs-CRP) | At Baseline and 12-week postintervention
  hs-CRP will be assessed using blood samples.
Changes of Adiponectin | At Baseline and 12-week postintervention
  Adiponectin will be assessed using blood samples.
Physical Function | At Baseline and 12-week postintervention
  Physical function, consisting of strength, flexibility, and agility components, will be assessed by the Senior's Fitness Test (SFT).
Health-Related Quality of Life | At baseline, 12-week (postintervention), 6-month, and 12-month
  Health-related quality of life will be assessed using the European Organization for Research and Treatment of Cancer- Quality of Life Questionnaire (EORTC-QLQ) - C30 questionnaire.
Prostate Cancer-Specific Quality of Life | At baseline, 12-week (postintervention), 6-month, and 12-month
  Prostate cancer-specific quality of life will be assessed using the Expanded Prostate Cancer Index Composite-26 (EPIC-26) questionnaire.
Fear of Cancer Progression | At baseline, 12-week (postintervention), 6-month, and 12-month
  Fear of cancer progression will be assessed using the Fear of Cancer Recurrence Inventory (FCRI) questionnaire.
Cancer Worry | At baseline, 12-week (postintervention), 6-month, and 12-month
  Cancer worry will be assessed using the Cancer Worry Scale (CWS) questionnaire.
General Anxiety | At baseline, 12-week (postintervention), 6-month, and 12-month
  General anxiety will be assessed using the Anxiety (general): Spielberger State-Trait Anxiety Inventory (STAI) questionnaire.
Prostate Cancer-Specific Anxiety | At baseline, 12-week (postintervention), 6-month, and 12-month
  Prostate cancer-specific anxiety will be assessed using the Memorial Anxiety Scale for Prostate Cancer (MAX-PC) questionnaire.
Depression | At baseline, 12-week (postintervention), 6-month, and 12-month
  Depression will be assessed using the Epidemiologic Studies Depression Scale (CES-D) questionnaire.
Perceived Stress | At baseline, 12-week (postintervention), 6-month, and 12-month
  Perceived stress will be assessed using the Perceived Stress Scale (PSS) questionnaire.
Self-esteem | At baseline, 12-week (postintervention), 6-month, and 12-month
  Self-esteem will be assessed using the Rosenberg Self-Esteem Scale (RSES) questionnaire.
Fatigue | At baseline, 12-week (postintervention), 6-month, and 12-month
  Fatigue will be assessed using the Functional Assessment of Cancer Therapy- Fatigue (FACT-F) questionnaire.
Physical Activity Level | At baseline, 12-week (postintervention), 6-month, and 12-month
  Physical activity level, consisting of light-, moderate-, and vigorous aerobic exercise and resistance exercise, will be assessed using the Godin Leisure-Time Exercise Questionnaire (GLTEQ).
Exercise Motivation | At baseline, 12-week (postintervention), 6-month, and 12-month
  Exercise motivation, consisting of Theory of Planned Behaviour (TPB) constructs (instrumental and affective attitudes, subjective norms, intention and perceived behavioral control), will be assessed using questionnaire.
Body composition | At baseline and 12-week (postintervention)
  Body composition, including body weight and waist- and hip-circumferences, will be assessed using weight scales and a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang DW, Fairey AS, Boule NG, Field CJ, Wharton SA, Courneya KS. Effects of Exercise on Cardiorespiratory Fitness and Biochemical Progression in Men With Localized Prostate Cancer Under Active Surveillance: The ERASE Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1487-1495. doi: 10.1001/jamaoncol.2021.3067. PMID 34410322
- [Result] Kang DW, Fairey AS, Boule NG, Field CJ, Wharton SA, Courneya KS. A Randomized Trial of the Effects of Exercise on Anxiety, Fear of Cancer Progression and Quality of Life in Prostate Cancer Patients on Active Surveillance. J Urol. 2022 Apr;207(4):814-822. doi: 10.1097/JU.0000000000002334. Epub 2022 Feb 17. PMID 35179044
- [Derived] Kang DW, Boule NG, Field CJ, Fairey AS, Courneya KS. Effects of supervised high-intensity interval training on motivational outcomes in men with prostate cancer undergoing active surveillance: results from a randomized controlled trial. Int J Behav Nutr Phys Act. 2022 Sep 29;19(1):126. doi: 10.1186/s12966-022-01365-2. PMID 36175907
- [Derived] Kang DW, Fairey AS, Boule NG, Field CJ, Courneya KS. Exercise duRing Active Surveillance for prostatE cancer-the ERASE trial: a study protocol of a phase II randomised controlled trial. BMJ Open. 2019 Jul 4;9(7):e026438. doi: 10.1136/bmjopen-2018-026438. PMID 31278095

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT03203460/Prot_SAP_000.pdf